CLINICAL TRIAL: NCT02400125
Title: China Cardiovascular Surgery Registry
Acronym: CCSR
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Collaborators: Ministry of Science and Technology of the People´s Republic of China (Other Government)
Responsible Party: Sponsor
Other Study IDs: MOST-2011BAI11B21; MOST-2011BAI11B02 (Other Grant/Funding Number: Ministry of Science and Technology of China)
Record Dates: First submitted 2015-03-22; First posted 2015-03-26 (Estimated); Last update posted 2015-12-16 (Estimated); Status verified 2015-12

CONDITIONS: Coronary Artery Bypass Grafting; Surgical Treatment for Heart Valve Diseases
Keywords: Patient Registry; Coronary Artery Bypass; Cardiac Valve Annuloplasty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 1: Patients underwent isolated or combined coronary artery bypass grafting surgery
- 2: Patients underwent isolate or combined surgical treatment for heart valve disease

SUMMARY:
China Cardiovascular Surgery Registry (CCSR) Study is a national database for coronary artery bypass grafting (CABG) and valve surgery performed in 87 hospitals with cardiovascular surgery volume > 100 per year. The aims of CCSR Study are: (i) report the characteristics of patient, the quality and evolvement of CABG and valve procedures in China, (ii) build and valid surgical risk assessment tools for Chinese population, (iii) provide databases for clinical studies, and quality improvement initiatives.

DETAILED DESCRIPTION:
The volume of cardiac surgery in China is increasing rapidly at a rate of approximately 10% annually, and has approached 207,881 at the year of 2013. Coronary artery bypass grafting (CABG) and valve procedures account for 41% of all. With the aging population, rising prevalence of cardiovascular diseases, and rapid economic development in China, the volume of cardiac procedures will continuously rise for years. In light of the burgeoning volume of cardiac procedures, considering the imbalance of economic development among regions, and the lack of standardized surgeon training system, critical concern with regards to the quality of cardiac surgery has been raised.

Under this circumstance, national registry to continuously collect patient-by-patient data for cardiovascular surgery is critically important to (i) report the characteristics of patient, the quality and evolvement of procedures, (ii) build and valid surgical risk assessment tools, (iii) provide databases for clinical studies, and quality improvement initiatives, (iv) promote international exchanges and cooperation. Following the example of national cardiac procedure databases, such as The Society of Thoracic Surgeons (STS) National Database and The European Association for Cardio-Thoracic Surgery (EACTS) Database, Fuwai Hospital, as one of the largest cardiac surgical care and research centers in China, leveraged an initiative to start the first multicenter cardiac surgery registry in Chinese mainland at 2004. The investigators started with 32 participating sites and registered CABG surgery during the first 2 years. From 2007, the investigators have included valve surgery as well. By the end of 2012, 66 coordinating sites have participated into this voluntary database continuously or intermittently, enrolled 61,558 surgery data. This database has become the most representative data source for adult cardiac surgery in China. This registry has (i) reported the performance and quality of adult cardiac surgery in China, shown that the observed and risk-adjusted in-hospital mortality rate of isolated CABG in China is 2.2% and 1.9% respectively, and identified certain variation among regions and sites, (ii) released an in-hospital mortality risk prediction system for CABG named SinoSCORE, which suit Chinese population better, (iii) worked with EACTS and merged both databases together for the 4th Adult Cardiac Surgical Database Report, (iv) acted as one platform and data source for clinical studies, published 14 papers in international indexed journals.

In order to extend the volume of participating sites, and build a representative database for the performance, in-hospital as well as 1-year outcomes of CABG and/or valve surgery in large cardiac surgery centers in China, at the year of 2013, China National Center for Cardiovascular Diseases (NCCD) and Fuwai Hospital leveraged The China Cardiovascular Surgery Registry (CCSR) network to push the CCSR Study forward. The CCSR Study established a network of 90 participating sites with cardiovascular surgery volume > 100 per year, and capability of performing CABG and/or valve surgery. The participating sites are required to consecutively and routinely submit CABG and valve surgery data regarding patients' personal information, risk factors, surgery performance, in-hospital outcomes and prescription drugs, through a web-based and paperless data collection system. The investigators also encourage all sites to interview patients at 1-month and 1-year after index procedure for mid-term outcomes and medications after discharge. The investigators conduct routine remote and on-site monitoring and auditing to ensure integrity and accuracy of data. Ethics Committee of Fuwai Hospital approved the study design and audits the conducting yearly.

For in-hospital data collection, CCSR established 11 modules (patient basic information, preoperative risks, cardiovascular presentation, cardiac examination, general information on operation, CABG, valve surgery, other surgeries, post-operative complications, pre-operative medication and medical order at discharge), 416 items, among which 157 items are core dataset, 259 are extended dataset. The core dataset is a mandatory set of variables believed to be necessary for accurate representation of clinical practice, risk model development, and analysis. The extended dataset includes less critical but still important fields that are strongly encouraged to be collected but are not mandatory for submitting. The creation of custom fields is permissible so that sites can collect specific information that is desired by themselves.

The investigators adapted Clinical Data Interchange Standards Consortium (CDISC) Standard for data collection and merging among international databases. The investigators established input items comparable to those of the STS National Database, the common terminologies and the definitions from STS National Database was adopted as well.

Coordinators are requested to consecutively register 5 variables regarding basic information of patients undergoing isolated or combined CABG and/or valve surgery in their hospital in 3 days after the surgery. The basic information includes name, sex, date of birth, type of surgery and ID number. The investigators request the coordinators to submit the complete in-hospital data within 28 days after the surgery. The investigators also developed a standard data interface for all in-hospital data elements. If the quality of participating sites' exported data from Hospital Information System meets the safety and quality criteria, it is also acceptable of these sites to export and import in-hospital data automatically instead of manual submitting.

The investigators encourage all participating sites to invite patients to join the prospective follow-up cohort and interview patients after discharge, but the follow-up interview is optional. Coordinators from participating sites interview the patients who have signed the informed consent during their index hospitalization and 1-month, 1-year after the index cardiac surgery face to face and by telephone. The data include major cardiovascular and cerebral outcomes, readmission, and self-administration.

In order to ensure the follow-up data authenticity, with the permission of patients and participating sites, NCC interviews patients at 3-month after their cardiac surgery using the same questionnaire.

Data variables have been added for internal quality and integrity checks. If any component of the required mandatory data elements are missing, or any of the validation roles of logic aren't meet, the data will be automatically rejected. In order to audit the accuracy of in-hospital data, the investigators randomly select 10-20% of each participating sites' in-hospital data, and require the coordinators to scan the coordinating medical record, and transferred to NCC using encryption flash drive. 2 physicians from NCC abstract all medical record data independently, and compare the data between NCC data abstraction and coordinators' database. The accuracy report of each sites are fed back to each participating site yearly. The on-site auditing are conducted once a year for each site. The main aim of on-site auditing is to ensure the consecutiveness of data registry. The investigators randomly select a period of time to check original record of surgery, and abstract data regarding patient ID and in-hospital outcomes. Any mismatch of auditing data with submitting data will be reported to NCC and participating sites.

ELIGIBILITY:
Inclusion Criteria:

* patients underwent isolated or combined coronary artery bypass grafting and/or surgical treatment for heart valve diseases

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients underwent isolated or combined coronary artery bypass grafting and/or surgical treatment for heart valve diseases
Sampling Method: Non-Probability Sample
Enrollment: 90000 (Estimated)
Dates: Start 2013-03; Primary Completion 2015-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
composite of post-operative all-cause mortality and major complications | participants will be followed for the duration of hospital stay after the index cardiac operation, an expected average of 2 weeks
  composite of death of any cause, reoperation, myocardial infarction, stroke, renal failure, pulmonary embolism, atrial fibrillation during the postoperative hospitalization

SECONDARY OUTCOMES:
major adverse cardiac events | 30 days
  composite of major adverse cardiac events (MACE) including death, myocardial infarction and/or revascularization
major adverse cardiac events | 1 year
  composite of major adverse cardiac events (MACE) including death, myocardial infarction and/or revascularization
readmission | 30 days
  composite of major adverse cardiac events (MACE) including death, myocardial infarction and/or revascularization
readmission | 1 year
  composite of major adverse cardiac events (MACE) including death, myocardial infarction and/or revascularization

CONTACTS AND LOCATIONS:
Overall Officials: Shengshou Hu, PhD, MD, Study Chair — Chinese Academy of Medical Sciences, Fuwai Hospital; Zhe Zheng, PhD, MD, Study Director — Chinese Academy of Medical Sciences, Fuwai Hospital
Locations (1):
- National Center for Cardiovascular Diseases, Fuwai Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Background] Deming Zhu CL, Feilong Hei. White Paper On 2013 China Cardiar Surgery And Extracorporeal Circulation Data. Chinese Journal of Extracorporeal Circulation 2014; 2014(3): 129-31.
- [Background] Shengshou Hu, Lingzhi Kong, Runlin Gao, et al. Report On Cardiovascular Diseases In China (2012). Encyclopedia of China Publishing House 2013.
- [Background] He J, Gu D, Wu X, Reynolds K, Duan X, Yao C, Wang J, Chen CS, Chen J, Wildman RP, Klag MJ, Whelton PK. Major causes of death among men and women in China. N Engl J Med. 2005 Sep 15;353(11):1124-34. doi: 10.1056/NEJMsa050467. PMID 16162883
- [Background] Moran A, Gu D, Zhao D, Coxson P, Wang YC, Chen CS, Liu J, Cheng J, Bibbins-Domingo K, Shen YM, He J, Goldman L. Future cardiovascular disease in china: markov model and risk factor scenario projections from the coronary heart disease policy model-china. Circ Cardiovasc Qual Outcomes. 2010 May;3(3):243-52. doi: 10.1161/CIRCOUTCOMES.109.910711. Epub 2010 May 4. PMID 20442213
- [Background] Yang G, Kong L, Zhao W, Wan X, Zhai Y, Chen LC, Koplan JP. Emergence of chronic non-communicable diseases in China. Lancet. 2008 Nov 8;372(9650):1697-705. doi: 10.1016/S0140-6736(08)61366-5. Epub 2008 Oct 17. PMID 18930526
- [Background] Wan YC, Wan YI. Delivering surgical training in the People's Republic of China: are current mechanisms adequate? Int J Surg. 2008 Dec;6(6):443-5. doi: 10.1016/j.ijsu.2008.08.012. Epub 2008 Sep 3. PMID 18838351
- [Background] Grover FL, Shahian DM, Clark RE, Edwards FH. The STS National Database. Ann Thorac Surg. 2014 Jan;97(1 Suppl):S48-54. doi: 10.1016/j.athoracsur.2013.10.015. No abstract available. PMID 24384250
- [Background] Head SJ, Howell NJ, Osnabrugge RL, Bridgewater B, Keogh BE, Kinsman R, Walton P, Gummert JF, Pagano D, Kappetein AP. The European Association for Cardio-Thoracic Surgery (EACTS) database: an introduction. Eur J Cardiothorac Surg. 2013 Sep;44(3):e175-80. doi: 10.1093/ejcts/ezt303. Epub 2013 Jun 19. PMID 23786918
- [Background] Zheng Z, Zhang L, Hu S, Li X, Yuan X, Gao H; Chinese Cardiovascular Surgical Registry Study. Risk factors and in-hospital mortality in Chinese patients undergoing coronary artery bypass grafting: analysis of a large multi-institutional Chinese database. J Thorac Cardiovasc Surg. 2012 Aug;144(2):355-9, 359.e1. doi: 10.1016/j.jtcvs.2011.10.012. Epub 2011 Nov 5. PMID 22056490
- [Background] Hu S, Zheng Z, Yuan X, Wang Y, Normand SL, Ross JS, Krumholz HM. Coronary artery bypass graft: contemporary heart surgery center performance in China. Circ Cardiovasc Qual Outcomes. 2012 Mar 1;5(2):214-21. doi: 10.1161/CIRCOUTCOMES.111.962365. Epub 2012 Mar 6. PMID 22396587
- [Background] Li Y, Zheng Z, Hu S; Chinese Coronary Artery Bypass Grafting Registry Study. The Chinese coronary artery bypass grafting registry study: analysis of the national multicentre database of 9248 patients. Heart. 2009 Jul;95(14):1140-4. doi: 10.1136/hrt.2008.146563. Epub 2008 Jul 16. PMID 18632834
- [Background] Zheng Z, Zhang L, Li X, Hu S; Chinese CABG Registry Study. SinoSCORE: a logistically derived additive prediction model for post-coronary artery bypass grafting in-hospital mortality in a Chinese population. Front Med. 2013 Dec;7(4):477-85. doi: 10.1007/s11684-013-0284-0. Epub 2013 Sep 18. PMID 24048813
- [Background] Zheng Z, Li Y, Zhang S, Hu S; Chinese CABG Registry Study. The Chinese coronary artery bypass grafting registry study: how well does the EuroSCORE predict operative risk for Chinese population? Eur J Cardiothorac Surg. 2009 Jan;35(1):54-8. doi: 10.1016/j.ejcts.2008.08.001. Epub 2008 Sep 7. PMID 18778949
- [Background] Zheng S, Zheng Z, Fan HG, Hu SS; Chinese Cardiovascular Surgery Registry. Is the European System for Cardiac Operative Risk Evaluation useful in Chinese patients undergoing heart valve surgery? Chin Med J (Engl). 2012 Oct;125(20):3624-8. PMID 23075714
- [Background] Ben Bridgewater RK, Jan Gummert, Peter Walton. Fourth EACTS Adult Cardiac Surgical Database Report: Towards Global Benchmarking. Dendrite Clinical Systems Limited 2010.
- [Background] Lamy A, Devereaux PJ, Prabhakaran D, Hu S, Piegas LS, Straka Z, Paolasso E, Taggart D, Lanas F, Akar AR, Jain A, Noiseux N, Ou Y, Chrolavicius S, Ng J, Yusuf S. Rationale and design of the coronary artery bypass grafting surgery off or on pump revascularization study: a large international randomized trial in cardiac surgery. Am Heart J. 2012 Jan;163(1):1-6. doi: 10.1016/j.ahj.2011.10.007. PMID 22172429
- [Derived] Wei Z, Zhu Z, Li Y, Li C, Liu N, Lu J, Wu M, Wang H, Xu D, Chen Y, Lai Y, Zhang H. Body Surface Area-Weighted Left Ventricular Ejection Fraction Enhances Prediction Accuracy of OPCABG Outcomes: A Large Multi-Center Cohort Study. Rev Cardiovasc Med. 2025 Nov 26;26(11):26681. doi: 10.31083/RCM26681. eCollection 2025 Nov. PMID 41356319
- [Derived] Zhu Z, Li Y, Zhang F, Steiger S, Guo C, Liu N, Lu J, Fan G, Wu W, Wu M, Wang H, Xu D, Chen Y, Zhu J, Meng X, Hou X, Anders HJ, Ye J, Zheng Z, Li C, Zhang H. Prediction of Male Coronary Artery Bypass Grafting Outcomes Using Body Surface Area Weighted Left Ventricular End-diastolic Diameter: Multicenter Retrospective Cohort Study. Interact J Med Res. 2023 Mar 23;12:e45898. doi: 10.2196/45898. PMID 36951893
- [Derived] Rao C, Zhang H, Gao H, Zhao Y, Yuan X, Hua K, Hu S, Zheng Z; Chinese Cardiac Surgery Registry Collaborative Group. The Chinese Cardiac Surgery Registry: Design and Data Audit. Ann Thorac Surg. 2016 Apr;101(4):1514-20. doi: 10.1016/j.athoracsur.2015.09.038. Epub 2015 Dec 1. PMID 26652141
- See also: the official website of Collaboration Association of Cardiovascular Surgeons in China — http://www.cvs-china.com/
- See also: login panel of China Cardiovascular Surgery Registry data up-sending and transmission system — http://ccsr.cvs-china.com/